CLINICAL TRIAL: NCT00570986
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of Two Dosing Regimens of ABT-874 to Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study Comparing the Safety and Efficacy of Two Dosing Regimens of ABT-874 to Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-890
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-01

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis
MeSH Terms: interventions — briakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Arm #1 is used for entire study. At week 12, arm is rerandomized.
  Interventions: Drug: Placebo
- 2 (Active Comparator): Arm #2 is used for entire study. At week 12, arm is rerandomized.
  Interventions: Biological: ABT-874
- 3 (Active Comparator): Arm #3 is not used for weeks 0-11. At week 12, arm is rerandomized.
  Interventions: Biological: ABT-874

INTERVENTIONS:
Drug: Placebo — Two injections at weeks 0 and 4. One injection at week 8. At week 12, arm is rerandomized to placebo every 4 weeks.
  Arms: 1
Biological: ABT-874 — 200mg at week 0 and week 4. 100mg at week 8. On week 12, arm is rerandomized to 100mg every 4 weeks.
  Arms: 2
Biological: ABT-874 — 100mg every 12 weeks.
  Arms: 3

SUMMARY:
The purpose of this study is to determine the safety and efficacy of 2 doses of ABT-874 versus placebo in the treatment of subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 18 years of age
* Subject had a clinical diagnosis of psoriasis for at least 6 months, and had moderate to severe plaque psoriasis
* Subject is judged to be in generally good health as determined by the principal investigator

Exclusion Criteria:

* Subject has previous exposure to systemic anti-IL 12 therapy
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid UVB or PUVA phototherapy
* Subject is taking or requires oral or injectible corticosteroids
* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, medication-induced or medication-exacerbated psoriasis or new onset guttate psoriasis
* Subject considered by the investigator, for any reason, to be an unsuitable candidate
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1465 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PGA | Proportion of subjects achieving a PGA 0/1 (Clear or minimal) at Week 12
PASI | Subjects achieving a PASI 75 response defined as a 75% reduction in the PASI score from baseline at Week 12
PGA | Proportion of subjects maintaining a PGA 0/1 response at Week 52

SECONDARY OUTCOMES:
DLQI | Change from Baseline in DLQI total score vs. placebo at Week 12
NAPSI | % change in NAPSI score at Week 12 vs placebo in subjects with nail psoriasis
PASI | Subjects who achieve PASI 90 and 100 at Week 12
Safety parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Chair — AbbVie
Locations (116):
- United States (93):
  - Site Reference ID/Investigator# 6579, Birmingham, Alabama
  - Site Reference ID/Investigator# 6697, Birmingham, Alabama
  - Site Reference ID/Investigator# 7015, Huntsville, Alabama
  - Site Reference ID/Investigator# 6728, Scottsdale, Arizona
  - Site Reference ID/Investigator# 6584, Tucson, Arizona
  - Site Reference ID/Investigator# 6696, Little Rock, Arkansas
  - Site Reference ID/Investigator# 6591, Bakersfield, California
  - Site Reference ID/Investigator# 6710, Fresno, California
  - Site Reference ID/Investigator# 7885, Irvine, California
  - Site Reference ID/Investigator# 6872, Los Angeles, California
  - Site Reference ID/Investigator# 7669, Oceanside, California
  - Site Reference ID/Investigator# 6821, San Diego, California
  - Site Reference ID/Investigator# 6832, San Diego, California
  - Site Reference ID/Investigator# 7305, San Diego, California
  - Site Reference ID/Investigator# 7990, San Francisco, California
  - Site Reference ID/Investigator# 6711, Santa Monica, California
  - Site Reference ID/Investigator# 8139, Torrance, California
  - Site Reference ID/Investigator# 7167, Vallejo, California
  - Site Reference ID/Investigator# 7302, Denver, Colorado
  - Site Reference ID/Investigator# 6921, Longmont, Colorado
  - Site Reference ID/Investigator# 6917, New Haven, Connecticut
  - Site Reference ID/Investigator# 6707, Jacksonville, Florida
  - Site Reference ID/Investigator# 7301, Miami, Florida
  - Site Reference ID/Investigator# 7012, Miami, Florida
  - Site Reference ID/Investigator# 6831, Miami, Florida
  - Site Reference ID/Investigator# 7016, South Miami, Florida
  - Site Reference ID/Investigator# 6590, West Palm Beach, Florida
  - Site Reference ID/Investigator# 6582, Alpharetta, Georgia
  - Site Reference ID/Investigator# 7450, Atlanta, Georgia
  - Site Reference ID/Investigator# 6714, Newnan, Georgia
  - Site Reference ID/Investigator# 6717, Snellville, Georgia
  - Site Reference ID/Investigator# 7017, Arlington Heights, Illinois
  - Site Reference ID/Investigator# 7877, Maywood, Illinois
  - Site Reference ID/Investigator# 6704, Skokie, Illinois
  - Site Reference ID/Investigator# 7292, West Dundee, Illinois
  - Site Reference ID/Investigator# 6706, Indianapolis, Indiana
  - Site Reference ID/Investigator# 7646, Indianapolis, Indiana
  - Site Reference ID/Investigator# 7014, Overland Park, Kansas
  - Site Reference ID/Investigator# 6873, Louisville, Kentucky
  - Site Reference ID/Investigator# 7523, Owensboro, Kentucky
  - Site Reference ID/Investigator# 6597, Andover, Massachusetts
  - Site Reference ID/Investigator# 6703, Boston, Massachusetts
  - Site Reference ID/Investigator# 7644, Detroit, Michigan
  - Site Reference ID/Investigator# 6826, Fort Gratiot, Michigan
  - Site Reference ID/Investigator# 7989, Grand Blanc, Michigan
  - Site Reference ID/Investigator# 6581, Fridley, Minnesota
  - Site Reference ID/Investigator# 7890, St Louis, Missouri
  - Site Reference ID/Investigator# 6709, St Louis, Missouri
  - Site Reference ID/Investigator# 7451, Omaha, Nebraska
  - Site Reference ID/Investigator# 7299, Berlin, New Jersey
  - Site Reference ID/Investigator# 6924, East Windsor, New Jersey
  - Site Reference ID/Investigator# 6577, New Brunswick, New Jersey
  - Site Reference ID/Investigator# 7030, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 7878, Buffalo, New York
  - Site Reference ID/Investigator# 7876, New York, New York
  - Site Reference ID/Investigator# 6599, New York, New York
  - Site Reference ID/Investigator# 6895, New York, New York
  - Site Reference ID/Investigator# 7637, New York, New York
  - Site Reference ID/Investigator# 7504, Rochester, New York
  - Site Reference ID/Investigator# 7018, Stoney Brook, New York
  - Site Reference ID/Investigator# 6926, Hickory, North Carolina
  - Site Reference ID/Investigator# 7293, Wilmington, North Carolina
  - Site Reference ID/Investigator# 8251, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 6598, Cincinnati, Ohio
  - Site Reference ID/Investigator# 8082, Cleveland, Ohio
  - Site Reference ID/Investigator# 7165, Columbus, Ohio
  - Site Reference ID/Investigator# 7659, Dayton, Ohio
  - Site Reference ID/Investigator# 6727, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 6894, Portland, Oregon
  - Site Reference ID/Investigator# 6578, Portland, Oregon
  - Site Reference ID/Investigator# 7295, Portland, Oregon
  - Site Reference ID/Investigator# 7879, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 6712, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6580, Johnston, Rhode Island
  - Site Reference ID/Investigator# 6576, Providence, Rhode Island
  - Site Reference ID/Investigator# 6589, Greer, South Carolina
  - Site Reference ID/Investigator# 6586, Goodlettsville, Tennessee
  - Site Reference ID/Investigator# 7668, Knoxville, Tennessee
  - Site Reference ID/Investigator# 6915, Nashville, Tennessee
  - Site Reference ID/Investigator# 6825, Arlington, Texas
  - Site Reference ID/Investigator# 6762, Austin, Texas
  - Site Reference ID/Investigator# 6822, Dallas, Texas
  - Site Reference ID/Investigator# 7671, Dallas, Texas
  - Site Reference ID/Investigator# 6705, Houston, Texas
  - Site Reference ID/Investigator# 6708, San Antonio, Texas
  - Site Reference ID/Investigator# 7081, San Antonio, Texas
  - Site Reference ID/Investigator# 6912, Tyler, Texas
  - Site Reference ID/Investigator# 7306, Webster, Texas
  - Site Reference ID/Investigator# 8101, Salt Lake City, Utah
  - Site Reference ID/Investigator# 6807, Norfolk, Virginia
  - Site Reference ID/Investigator# 6801, Seattle, Washington
  - Site Reference ID/Investigator# 7519, Spokane, Washington
  - Site Reference ID/Investigator# 7080, Milwaukee, Wisconsin
- Canada (23):
  - Site Reference ID/Investigator# 7314, Barrie
  - Site Reference ID/Investigator# 7452, Calgary
  - Site Reference ID/Investigator# 6702, Edmonton
  - Site Reference ID/Investigator# 6716, Halifax
  - Site Reference ID/Investigator# 7309, Hamilton
  - Site Reference ID/Investigator# 6588, Laval
  - Site Reference ID/Investigator# 6715, London
  - Site Reference ID/Investigator# 7315, London
  - Site Reference ID/Investigator# 7636, Markham
  - Site Reference ID/Investigator# 6699, Montreal
  - Site Reference ID/Investigator# 7316, Montreal
  - Site Reference ID/Investigator# 7088, North Bay
  - Site Reference ID/Investigator# 7310, Ottawa
  - Site Reference ID/Investigator# 7311, Québec
  - Site Reference ID/Investigator# 7313, St. John's
  - Site Reference ID/Investigator# 7317, Surrey
  - Site Reference ID/Investigator# 7308, Vancouver
  - Site Reference ID/Investigator# 6713, Vancouver
  - Site Reference ID/Investigator# 7067, Waterloo
  - Site Reference ID/Investigator# 7312, Westmount
  - Site Reference ID/Investigator# 7087, Windsor
  - Site Reference ID/Investigator# 6805, Windsor
  - Site Reference ID/Investigator# 7638, Winnipeg